CLINICAL TRIAL: NCT00360711
Title: Genetic Counselors' Experiences of Moral Value Conflicts With Clients
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906179; 06-HG-N179
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-31

CONDITIONS: Moral Value Conflicts; Moral Distress; Genetic Counseling
Keywords: Moral Distress; Nondirectiveness; Ethical Dilemma

SUMMARY:
This study will examine the experience of moral value conflicts among genetic counselors. Previous research has shown that value conflicts do exist among genetic counselors, but little is known about the nature or consequences of these conflicts. This is a sub-study of the "Manifestations and Consequences of Moral Distress Among Genetic Service Providers: An Exploratory Study," which includes genetic counselors, nurses and medical geneticists.

Genetic counselors are recruited for this value-conflict sub-study from among those participating in the Moral Distress study. Participants are interviewed in-depth by telephone about their experiences of moral value conflicts with clients. The interviews cover the following: situations in which the counselor has disagreed with a client's decision or views on a moral level; the counselor's thought processes during and after a session in which conflicts arise; the counselor's feelings and emotions associated with sessions involving a moral value conflict; the counselor's current and previous work settings; the counselor's view of his or her role and responsibility in a client's decision; challenging a client's values or decision; and preparation for value conflicts.

DETAILED DESCRIPTION:
Genetic counselors may be faced with situations in which they disagree on a moral level with the views or decisions of their clients. These moral value conflicts between counselors and their clients may have negative emotional consequences for counselors. Little is known about the range of sources of these conflicts, the approaches counselors take to address them, or the impact they have on the counselor's life and career. This study seeks to gain insight into the nature, sources, and consequences of moral value conflicts among genetic counselors through semi-structured in-depth interviews with approximately 30 genetic counselors. Interview questions will be nested within interviews for a larger study entitled "Moral Distress and Suffering of Genetics Professionals". The discussion will be centered on a personal experience of moral value conflict that the counselor has had with a client. Interviews will be transcribed and subjected to thematic analysis. Such analysis will result in the identification of common themes running through the interviews. An understanding of value conflicts may allow for future interventions to minimize the negative effects of these events.

ELIGIBILITY:
* INCLUSION / EXCLUSION CRITERIA:

A sample of approximately 30 genetic counselors will be interviewed for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Start 2006-06-01; Study Completion 2007-03-31

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Hodgson J, Spriggs M. A practical account of autonomy: why genetic counseling is especially well suited to the facilitation of informed autonomous decision making. J Genet Couns. 2005 Apr;14(2):89-97. doi: 10.1007/s10897-005-4067-x. PMID 15959640